CLINICAL TRIAL: NCT02004210
Title: A Randomized, Multi-center, Open Label, Phase 3 Trial Comparing Conventional TACE and Transarterial Radioembolization in Patients With Unilobar Advanced Hepatocellular Carcinoma
Brief Title: A Phase 3 Trial Comparing TACE and TARE in Unilobar Advanced Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participants were enrolled.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Hwan Yoon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACE_TARE
Record Dates: First submitted 2013-10-01; First posted 2013-12-09 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: transarterial chemoembolization; transarterial radioembolization; advanced hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The TARE group (Experimental): transarterial radioembolization group
  Interventions: Procedure: transarterial radioembolization (TARE)
- The TACE group (Experimental): Transarterial chemoembolization group
  Interventions: Procedure: transarterial chemoembolization (TACE)

INTERVENTIONS:
Procedure: transarterial radioembolization (TARE) — transarterial radioembolization
  Arms: The TARE group
Procedure: transarterial chemoembolization (TACE) — transarterial chemoembolization
  Arms: The TACE group

SUMMARY:
The aim of this study is to compare the efficacy of conventional transarterial chemoembolization(TACE) and transarterial radioembolization in patients with unilobar advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Potentially curative treatments for hepatocellular carcinoma (HCC) include surgical resection, liver transplantation, and local ablative therapy.

However, HCC patients are diagnosed at advanced stages in Korea. Unresectable advanced HCCs are not suitable for other curative therapies. For these patients, the optimal treatment remains largely controversial. As a palliative treatment, the benefit of transarterial chemoembolization (TACE) had been shown in patients with unresectable HCC by several trials. Recently,transarterial radioembolization (TARE) has been introduced for the treatment of advanced HCC. However, the efficacy of TARE compared to TACE is uncertain.

The aim of this study is to compare the efficacy of conventional transarterial chemoembolization(TACE) and transarterial radioembolization in patients with unilobar advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical or histological diagnosis of HCC based on the guidelines of the AJCC
* Patients with advanced HCC with unilobar advanaced involvement: right lobe ± S4 segment or left lobe ± S4 segment)
* Patients with single large HCC or multinodular HCC

  * Single & 5cm < size < 15cm
  * 2-5 nodules & maximal sized 4-15cm & sum of diameters ≦ 25cm
  * Infiltrative type & unilobular involvement on liver MRI
  * Segmental or lobar portal vein invasion can be included.
* Age : 20 years to 80 years
* ECOG Performance Status of 0 to 2
* Child-Pugh class A (Child-Pugh score 5-6), B (CP score 7)
* Adequate bone marrow, liver function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * WBC count ≧ 1,000/mm3
  * Absolute neutrophil count > 500/mm3
  * Hb ≧ 7.0 g/dL
  * Platelet count > 100,000 /mm3
  * Bilirubin ≦ 3 mg/dL
  * Adequate clotting function: INR ≦ 2.3 or ≦ 6sec

Exclusion Criteria:

* Child-Pugh score ≧ 8
* ECOG Performance Status ≧ 3
* Patients with chronic kidney disease or serum creatinine ≥ 1.2 mg/dL
* History of organ allograft
* Patients with uncontrolled co-morbidity which needs treatment
* Patients who have received prior systemic chemotherapy
* Patients who have received Capecitabine within 8 weeks
* Patients with extrahepatic metastasis
* Main portal vein invasion
* Patients with lymph node metastasis
* Bilobar involvement
* Bulk disease(Tumor volume >70% of the target liver volume, or tumor nodules too numerous to count)
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | every 12 weeks, up to the time of death, up to 12 months
  From date of randomization until the date of death

SECONDARY OUTCOMES:
Progression-Free Survival in the Liver | every 12 weeks, up to the time of death or first documented intrahepatic tumor progression, up to 12 months
  From date of randomization until the date of first documented intrahepatic tumor progression or death
Progression-Free Survival Overall | every 12 weeks, up to the time of death or first documented progression, up to 12 months
  From date of randomization until the date of first documented progression or death
Overall tumor response assessment | every 12 weeks, up to the time of death or 12 months
  (CR, PR, SD, PD)by modified RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hwan Yoon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea